CLINICAL TRIAL: NCT02855996
Title: Evaluation of AVANCE Fathers in Action/Padres Activos Fatherhood Program
Acronym: AVANCE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: AVANCE (Grantee and Implementing Agency) relinquished funding. Subsequently, both program and evaluation were terminated prematurely.
Sponsor: University of Texas at Austin (Other)
Responsible Party: Principal Investigator, Cynthia Osborne, Faculty/Rsearcher, Associate Professor, University of Texas at Austin
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AVANCE
Record Dates: First submitted 2016-07-28; First posted 2016-08-04 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Fathers
Keywords: fatherhood; father involvement; economic stability; co-parenting; healthy relationships; father-child engagement

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Fathers will be randomly assigned to participate in the "Fathers in Action/Padres Activos (FA/PA)" intervention program to support fathers' healthy relationships with their children and support their co-parenting skills.
  Interventions: Other: Fathers in Action/Padres Activos (FA/PA) program
- Control (No Intervention): Fathers waitlisted for participation in the "Fathers in Action/Padres Activos (FA/PA)" program.

INTERVENTIONS:
Other: Fathers in Action/Padres Activos (FA/PA) program — The program focuses on increasing the father's role in the child's education, nurturing and bonding with the child, loving and respecting the child's mother, coaching the child, and serving as a role model. The program also includes employment coaching.
  Other Names: FA/PA program
  Arms: Intervention

SUMMARY:
The Child and Family Research Partnership (CFRP) will be conducting the "local" evaluation of AVANCE's Fathers in Action/Padres Activos (FA/PA) fatherhood program. AVANCE is a non-profit organization that has served low-income families and children since its founding in 1973. AVANCE sites have been providing fatherhood services for some time, but the programming offered has varied across sites and no rigorous evaluation of the programs has been completed. Through a federally-funded Responsible Fatherhood grant, AVANCE aims to create one fatherhood curriculum to be used across their sites: Fathers in Action/Padres Activos (FA/PA).

The purpose of the study is to advance the field of knowledge in the area of fatherhood programing by providing rigorous evidence on the impact of a comprehensive fatherhood program on enhancing a father's ability to be involved with and parent his child, in addition to providing more information on the selective characteristics of fathers who choose to participate in fatherhood programs. The study will seek to answer the following research questions: (1) What are the demographic and relationship characteristics of fathers who choose to participate in the Fathers in Action/Padres Actívos (FA/PA) program, and how do these characteristics compare to the fathers associated with mothers and children in other AVANCE programs?; (2) Does the FA/PA program positively impact parenting and co-parenting, father engagement and involvement, and healthy relationship?; (3) Are the program impacts similar for low-income fathers across regions (Houston v. the Rio Grande Valley), race/ethnicity (African American v. Hispanic), and coresidential status (nonresident v. resident)?; and (4) What are the factors that enhance or impede the successful implementation of the FA/PA program?

ELIGIBILITY:
Inclusion Criteria:

* Fathers (biological, adoptive, or social) over 18 years of age
* Able to travel to program location to attend classes

Exclusion Criteria:

* Under 18 years of age
* Female

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-09 (Actual)

PRIMARY OUTCOMES:
Number of fathers reporting healthy father-child involvement and bond | Six months
  Increase healthy father-child involvement and bond (connectedness) among residential and non-residential fathers of children 0-5 years. Scale of items (never - often) aggregated to create a score on the outcome. Will report number of treatment fathers whose score is higher than control group fathers at 6 months.
Number of fathers reporting healthy co-parenting relationship | Six months
  Establish and maintain healthy co-parenting relationship among residential and non-residential fathers of children 0-5 years. Scale of items (never - always) aggregated to create a score on the outcome. Will report number of treatment fathers whose score is higher than control group fathers at 6 months.
Number of fathers reporting development of "self as father" | Six months
  Strengthen the development of "self as father" among residential and non-residential fathers of children 0-5 years. Several items (anger and stress management, financial stability, personal development) aggregated to create a score on the outcome. Will report number of treatment fathers whose score is higher than control group fathers at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Cynthia Osborne, PhD, Principal Investigator — University of Texas at Austin

IPD SHARING:
Plan to Share IPD: No